CLINICAL TRIAL: NCT04734418
Title: Evaluation of Remifentanil and Dexmedetomidine in Patients With Noninvasive Mechanical Ventilation Intolerance After Cardiac Surgery: a Multicenter, Prospective, Single-blind, Randomized Controlled Study
Brief Title: Evaluation of Remifentanil and Dexmedetomidine in Patients With Noninvasive Mechanical Ventilation Intolerance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Guowei Tu, Associated professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REDNIVI
Record Dates: First submitted 2021-01-22; First posted 2021-02-02 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: NIV Intolerance
MeSH Terms: interventions — Remifentanil; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remifentanil group (Experimental)
  Interventions: Drug: Remifentanil
- Dexmedetomidine (Active Comparator)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Remifentanil — Intravenous pump injection.The initial dose of remifentanil is 0.05 μg/kg/min.The drug dosage will be adjusted according to the subjects' intolerance relief (the treatment target is NIS ≤ 2), and the maximum dosage of remifentanil is 0.12 μg/kg/min
  Arms: Remifentanil group
Drug: Dexmedetomidine — Intravenous pump injection.The initial dose of dexmedetomidine is 0.5 μg/kg/h.The drug dosage will be adjusted according to the subjects' intolerance relief (the treatment target is NIS ≤ 2), and the maximum dosage of dexmedetomidine is 1.0 μg/kg/h.
  Arms: Dexmedetomidine

SUMMARY:
Currently, NIV(Noninvasive ventilation ) is widely used in patients with hypoxemia and atelectasis after cardiac surgery.About 15% of patients have intolerance during NIV. The main manifestation is that the patient feels uncomfortable, often breaks away from the mask, and even gradually becomes agitated, which eventually leads to the failure of non-invasive ventilation.The patient's intubation rate is as high as 44%, and the mortality rate is 34%.There are many ways to prevent or treat NIV intolerance, of which the most used is to sedate the patient. This study aims to evaluate the effects of remifentanil and dexmedetomidine in the sedation of patients with intolerance to non-invasive mechanical ventilation after cardiac surgery, and to explore the optimal plan for sedation of patients with intolerant non-invasive mechanical ventilation after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form voluntarily and follow the plan requirements;
* Age from 18 to 75 years old (including 18 and 75 years old), regardless of gender;
* Patients who received non-invasive mechanical ventilation after cardiac surgery and were intolerant of non-invasive ventilation.

Exclusion Criteria:

* A history of allergy to any component of the study drug;
* Visual analogue scale of pain (VAS) score >4；
* Who had taken dexmedetomidine within 8 hours prior to the study;
* Who had used remifentanil within 2 hours before the study began;
* Expectoration difficulties;
* Women who are pregnant or lactating;
* Coma or uncontrollable convulsions;
* Have a history of mental illness or cognitive impairment;
* Delirium before the study began;
* Patients with severe liver dysfunction (CTP grade C);
* Patients with renal insufficiency (patients receiving renal replacement therapy);
* Preoperative left ventricular ejection fraction (LVEF) < 30%;
* History of drug and alcohol abuse;
* Other conditions that the investigator deems inappropriate for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Remission rate of intolerance in patients with intolerance of non-invasive mechanical ventilation after cardiac surgery after sedation with remifentanil or dexmedetomidine. | Within 72 hours of study drug used

SECONDARY OUTCOMES:
Mortality in both remifentanil and dexmedetomidine group | Up to 30 days
Mechanical ventilation time in both remifentanil and dexmedetomidine group | Up to 30 days
Hemodynamic changes in both remifentanil and dexmedetomidine group | Up to 30 days
Incidence of delirium in both remifentanil and dexmedetomidine group | Up to 30 days
Days in ICU in both remifentanil and dexmedetomidine group | Up to 30 days
Intubation rate in both remifentanil and dexmedetomidine group | Up to 30 days
Tracheotomy rate in both remifentanil and dexmedetomidine group | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Luo, MD PhD, Study Chair — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Hao GW, Luo JC, Xue Y, Ma GG, Su Y, Hou JY, Yu SJ, Liu K, Zheng JL, Tu GW, Luo Z. Remifentanil versus dexmedetomidine for treatment of cardiac surgery patients with moderate to severe noninvasive ventilation intolerance (REDNIVIN): a prospective, cohort study. J Thorac Dis. 2020 Oct;12(10):5857-5868. doi: 10.21037/jtd-20-1678. PMID 33209418
- [Derived] Hao GW, Wu JQ, Yu SJ, Liu K, Xue Y, Gong Q, Xie RC, Ma GG, Su Y, Hou JY, Zhang YJ, Liu WJ, Li W, Tu GW, Luo Z. Remifentanil vs. dexmedetomidine for cardiac surgery patients with noninvasive ventilation intolerance: a multicenter randomized controlled trial. J Intensive Care. 2024 Sep 18;12(1):35. doi: 10.1186/s40560-024-00750-2. PMID 39294818
- [Derived] Deng YZ, Luo MH, Luo JC, Li JK, Chen JQ, Zhang YJ, Hou JY, Su Y, Tu GW, Luo Z. Postoperative glucocorticoids in patients with acute type A aortic dissection (GLAD): study protocol for a prospective, single-center, randomized controlled trial. BMC Anesthesiol. 2023 May 15;23(1):164. doi: 10.1186/s12871-023-02124-x. PMID 37189085
- [Derived] Luo MH, Hao GW, Liu K, Yin K, Yu SJ, Wang H, Su Y, Luo JC, Wei YQ, Wang YH, Pan WQ, Tu GW, Luo Z. Remifentanil versus Dexmedetomidine in Cardiac Surgery Patients with Noninvasive Ventilation Intolerance: Protocol for the REDNIVI Trial. Rev Cardiovasc Med. 2022 Mar 4;23(3):84. doi: 10.31083/j.rcm2303084. PMID 35345251
- See also: Remifentanil versus dexmedetomidine for treatment of cardiac surgery patients with moderate to severe noninvasive ventilation intolerance (REDNIVIN): a prospective, cohort study — https://jtd.amegroups.com/article/view/44501/html